CLINICAL TRIAL: NCT01244529
Title: Comparison of Lens Fit and Lens Power of a New Contact Lens to Two Marketed Contact Lenses in a Population of Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CR-201011
Record Dates: First submitted 2010-11-17; First posted 2010-11-19 (Estimated); Results first posted 2012-01-24 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2017-08

CONDITIONS: Myopia
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- galy A Plus/ galy A / seno A (Other): Pair 1: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 2: galy A-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 3: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A
- galy A Plus / seno A / galy A (Other): Pair 1: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 2: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Pair 3: galy A-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A
- galy A / galy A Plus / seno A (Other): Pair 1: galy A-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 2: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 3: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A
- galy A / seno A / galy A Plus (Other): Pair 1: galy A-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 2: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Pair 3: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A
- seno A / galy A / glay A Plus (Other): Pair 1: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Pair 2: galy A-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 3: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A
- seno A / galy A Plus / galy A (Other): Pair 1: seno A- subjects were randomized to receive different base curves for each eye (BC: 8.4 or 8.8).
  Pair 2: galy A Plus-subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Pair 3: galy A -subjects were randomized to receive different base curves for each eye (BC: 8.3 or 8.7).
  Interventions: Device: galy A Plus; Device: seno A; Device: galy A

INTERVENTIONS:
Device: galy A Plus — galyfilcon A Plus, BC: 8.3 or 8.7
Device: seno A — senofilcon A, BC:8.4 or 8.8
Device: galy A — galyfilcon A , BC: 8.3 or 8.7

SUMMARY:
The purpose of this study is to evaluate the comparability of lens fit and lens power of a new contact lens to the lens fit and lens power of two marketed lenses.

ELIGIBILITY:
Inclusion Criteria:

* Must be at least 18 years of age and no more than 55 years of age.
* Must sign written informed consent.
* Optimal spherical equivalent distance correction must be between -1.00 and -6.00 diopters.
* Have spectacle astigmatism ≤ -0.75 diopter cylinder in both eyes.
* Must have visual acuity best correctable to 20/25+3 or better for each eye.
* Must appear able and willing to adhere to the instructions set forth in this clinical protocol.
* Have normal eyes with no evidence of abnormality or disease. For the purposes of this study a normal eye is defined as one having: No evidence of lid abnormality or infection; No conjunctival abnormality or infection; No clinical significant slit lamp findings, (i.e., oedema, staining, scarring, vascularization, infiltrates or abnormal opacities); No other active ocular disease.
* The subject is a current spherical soft contact lens wearer (defined as a minimum of 6 hours of daily wear for a minimum of 1 month prior to the study) and willing to wear the study lenses on a daily wear basis (defined as a minimum of 6 hours of wear per day at least five days of the week) for the duration of the study.

Exclusion Criteria:

* Any systemic illness which would contraindicate lens wear or the medical treatment of which would affect vision or successful lens wear.
* Any previous eye surgery involving the anterior segment.
* Pre-existing ocular disease that would preclude contact lens fitting.
* Abnormal lacrimal secretions.
* Keratoconus or other corneal irregularity.
* Pregnancy, lactating or planning a pregnancy at the time of enrollment.
* Participation in any concurrent clinical trial.
* Subject's habitual contact lens type is toric or multifocal.
* Require any concurrent ocular medication.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2010-09-01 (Actual); Primary Completion 2010-11-01 (Actual); Study Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - Farnham, Surrey
  - Birmingham

RESULTS

PARTICIPANT FLOW:
Groups:
- All Arms, All Interventions: All subjects wore all intervention throughout the course of the study.
Period: Overall Study
Arm/Group | All Arms, All Interventions
Started | 41
Completed | 41
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled subjects.
Groups:
- All Subjects: All subjects who where enrolled wore all intervention lenses throughout the course of the study. The specific lenses used include the following: senofilcon A (control) soft contact lens with 8.8 base; senofilcon A (control) soft contact lens with 8.4 base curve; galyfilcon A (control) soft contact lens with 8.7 base curve; galyfilcon A (control) soft contact lens with 8.3 base curve; galyfilcon A Plus (test) soft contact lens with 8.7 base curve; galyfilcon A Plus (test) soft contact lens with 8.3 base curve.
Arm/Group | All Subjects
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 20
Region of Enrollment [Number; unit: participants]
  United Kingdom | 41

OUTCOME MEASURES:

1. Primary Outcome: Lens Centration Acceptance
Description: Investigator evaluated as acceptable (centered/slightly decentered) or unacceptable (substantially decentered). Number of eyes in each category will be reported by lens. This is an aggregate reporting of the lenses, combining the different base curves into a category by lens type. This is done per protocol, due to this primary outcome not being stratified by base curve.
Time Frame: after 15 minutes of contact lens wear
Population: Analysis was on those completed subjects who were enrolled, randomized, and assigned to a study arm.
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Groups:
- Galyfilcon A Plus (Test); Galyfilcon A (Control); Senofilcon A: All subjects wore each of the lenses at a point in the study as this was a contralateral study.
Arm/Group | Galyfilcon A Plus (Test) | Galyfilcon A (Control) | Senofilcon A
Number analyzed (Participants) | 41 | 41 | 41
Number analyzed (eyes) | 82 | 82 | 82
eyes
  Acceptable centration | 74 | 62 | 69
  Unacceptable centration | 8 | 20 | 13

2. Primary Outcome: Primary Gaze Lens Movement
Description: Investigator evaluated as acceptable (minimal or moderate movement) or unacceptable (insufficient or excessive movement). Percent of eyes in each category will be evaluated.
Time Frame: after 15 minutes of contact lens wear
Population: Analysis was on those completed subjects who were enrolled, randomized, and assigned to a study arm.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Galyfilcon AP 8.3 BC; Galyfilcon A 8.3 BC; Senofilcon A 8.4 BC; Galyfilcon AP 8.7 BC; Galyfilcon A 8.7 BC; Senofilcon A 8.8 BC: All subjects wore each of the lenses at a point in the study as this was a contralateral study.
Arm/Group | Galyfilcon AP 8.3 BC | Galyfilcon A 8.3 BC | Senofilcon A 8.4 BC | Galyfilcon AP 8.7 BC | Galyfilcon A 8.7 BC | Senofilcon A 8.8 BC
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41 | 41
Number analyzed (eyes) | 41 | 41 | 41 | 41 | 41 | 41
percentage of eyes
  Acceptable movement | 93 | 93 | 100 | 93 | 90 | 98
  Unacceptable movement | 7 | 7 | 0 | 7 | 10 | 2

3. Primary Outcome: Fit Acceptability
Description: Investigator evaluated lens fit using a six point scale: 5-optimal...3-borderline acceptable...2-unacceptable. Percent of eyes in each category will be evaluated.
Time Frame: after 15 minutes of contact lens wear
Population: Analysis was on those completed subjects who were enrolled, randomized, and assigned to a study arm.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Arm/Group | Galyfilcon AP 8.3 BC | Galyfilcon A 8.3 BC | Senofilcon A 8.4 BC | Galyfilcon AP 8.7 BC | Galyfilcon A 8.7 BC | Senofilcon A 8.8 BC
Number analyzed (Participants) | 41 | 41 | 41 | 41 | 41 | 41
Number analyzed (eyes) | 41 | 41 | 41 | 41 | 41 | 41
percentage of eyes
  Acceptable Fit | 90 | 90 | 95 | 83 | 71 | 80
  Unacceptable Fit | 10 | 10 | 5 | 17 | 29 | 20

4. Secondary Outcome: New Lens Power Fit Match to Control Lenses
Description: The lens power fit of test lenses will be compared to control lenses to determine if the power matches. Percent of eyes with exact power fit will be evaluated.
Time Frame: after 15 minutes of contact lens wear
Population: Analysis was on those completed subjects who were enrolled, randomized, and assigned to a study arm.
Measure: Number; unit: percentage of eyes
Units Other Than Participants: eyes
Groups:
- Galyfilcon AP 8.3 BC vs Galyfilcon A 8.3 BC; Galyfilcon AP 8.3 BC vs Senofilcon A 8.4 BC; Galyfilcon AP 8.7 BC vs Galyfilcon A 8.7 BC; Galyfilcon AP 8.7 BC vs Senofilcon A 8.8 BC: All subjects wore each of the lenses at a point in the study as this was a contralateral study.
Arm/Group | Galyfilcon AP 8.3 BC vs Galyfilcon A 8.3 BC | Galyfilcon AP 8.3 BC vs Senofilcon A 8.4 BC | Galyfilcon AP 8.7 BC vs Galyfilcon A 8.7 BC | Galyfilcon AP 8.7 BC vs Senofilcon A 8.8 BC
Number analyzed (Participants) | 41 | 41 | 41 | 41
Number analyzed (eyes) | 41 | 41 | 41 | 41
percentage of eyes
  Lens Power the Same | 98 | 98 | 98 | 98
  Lens Power Not the Same | 2 | 2 | 2 | 2

ADVERSE EVENTS:
Arm/Group | All Arms, All Interventions
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires agreement and written authorization from Sponsor.